CLINICAL TRIAL: NCT07071753
Title: OPT-FRESH: Optimizing Online Purchasing of Fruits, Vegetables, and Legumes for Low-Income Families
Brief Title: Optimizing Online Purchasing of Fruits, Vegetables, and Legumes for Low-Income Families
Acronym: OPT-FRESH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-FY2025-10110
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Food Insecurity; Healthy Eating
Keywords: MOST; Healthy eating; Online grocery purchase; SNAP

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Texting + Financial Incentive + Shoppable List (Experimental): Online grocer delivery fee waiver and a tutorial video addressing digital literacy will be constant components, meaning that it will be available to all participants in the study. Plus:
  1. weekly text messages to improve the trust in online grocery services;
  2. weekly match-up to $10 as a financial incentive for purchasing FVL online targeting loss aversion;
  3. weekly instant shoppable grocery lists of culturally tailored meal suggestions using SNAP recipes targeted at impulse purchases.
  Interventions: Behavioral: Video tutorial; Behavioral: Delivery fee waiver; Behavioral: Texting; Behavioral: Financial incentive; Behavioral: Grocery list with instant shoppable SNAP-Ed recipes
- Texting + Financial Incentive (Experimental): Online grocer delivery fee waiver and a tutorial video addressing digital literacy will be constant components, meaning that it will be available to all participants in the study. Plus:
  1. weekly text messages to improve the trust in online grocery services;
  2. weekly match-up to $10 as a financial incentive for purchasing FVL online targeting loss aversion;
  Interventions: Behavioral: Video tutorial; Behavioral: Delivery fee waiver; Behavioral: Texting; Behavioral: Financial incentive
- Texting only (Experimental): Online grocer delivery fee waiver and a tutorial video addressing digital literacy will be constant components, meaning that it will be available to all participants in the study. Plus:
  1) weekly text messages to improve the trust in online grocery services;
  Interventions: Behavioral: Video tutorial; Behavioral: Texting
- Financial Incentive + Shoppable List (Experimental): Online grocer delivery fee waiver and a tutorial video addressing digital literacy will be constant components, meaning that it will be available to all participants in the study. Plus:
  1. weekly match-up to $10 as a financial incentive for purchasing FVL online targeting loss aversion;
  2. weekly instant shoppable grocery lists of culturally tailored meal suggestions using SNAP recipes targeted at impulse purchases.
  Interventions: Behavioral: Video tutorial; Behavioral: Delivery fee waiver; Behavioral: Financial incentive; Behavioral: Grocery list with instant shoppable SNAP-Ed recipes
- Texting + Shoppable List (Experimental): Online grocer delivery fee waiver and a tutorial video addressing digital literacy will be constant components, meaning that it will be available to all participants in the study. Plus:
  1. weekly text messages to improve the trust in online grocery services;
  2. weekly instant shoppable grocery lists of culturally tailored meal suggestions using SNAP recipes targeted at impulse purchases.
  Interventions: Behavioral: Video tutorial; Behavioral: Delivery fee waiver; Behavioral: Texting; Behavioral: Grocery list with instant shoppable SNAP-Ed recipes
- Shoppable List (Experimental): Online grocer delivery fee waiver and a tutorial video addressing digital literacy will be constant components, meaning that it will be available to all participants in the study. Plus:
  1) weekly instant shoppable grocery lists of culturally tailored meal suggestions using SNAP recipes targeted at impulse purchases.
  Interventions: Behavioral: Video tutorial; Behavioral: Delivery fee waiver; Behavioral: Grocery list with instant shoppable SNAP-Ed recipes
- Financial Incentive (Experimental): Online grocer delivery fee waiver and a tutorial video addressing digital literacy will be constant components, meaning that it will be available to all participants in the study. Plus:
  1) weekly match-up to $10 as a financial incentive for purchasing FVL online targeting loss aversion.
  Interventions: Behavioral: Video tutorial; Behavioral: Delivery fee waiver; Behavioral: Financial incentive
- Delivery fee waived only (Active Comparator): Online grocer delivery fee waiver and a tutorial video addressing digital literacy will be constant components, meaning that it will be available to all participants in the study.
  Interventions: Behavioral: Video tutorial; Behavioral: Delivery fee waiver

INTERVENTIONS:
Behavioral: Video tutorial — At the onset of the intervention, all participants will receive tutorial videos via text, covering Instacart account setup, online item selection, and SNAP-eligible stores, aiming to improve digital literacy in grocery shopping. The video was developed by our team, reviewed by SNAP-Ed partners, and available in English and Spanish. Despite being considered helpful during the pilot, nearly half of the participants reported not receiving or watching the tutorial video. To address this, we will call all participants within the trial's first week to provide technical assistance, including step-by-step instructions on redemption of the free delivery membership. Phone follow-ups were well-received during the pilot. Also, an intervention package will be mailed to all participants as material to be referred to in the calls and throughout the intervention. Those receiving the grocery list component will receive shopping lists and recipes printed and via SMS, to aid online grocery ordering in si
Behavioral: Delivery fee waiver — All participants will receive a 12-week Instacart+ Membership e-gift card, eliminating the online delivery fee for orders >$35.
  Arms: Delivery fee waived only; Financial Incentive; Financial Incentive + Shoppable List; Shoppable List; Texting + Financial Incentive; Texting + Financial Incentive + Shoppable List; Texting + Shoppable List
Behavioral: Texting — Participants randomized to this component will receive 2 text messages weekly via EZ text to enhance their perception of behavioral control and trust in online grocery services. Text messages, deemed acceptable during our pilot, will be actionable, informed by constructs of the Theory of Planned Behavior, and tailored to assist shoppers using Instacart delivery services. We will deliver 24 short text messages (<160 characters), on Friday afternoons and Mondays, each with one or more of the purposes rooted in behavior change techniques: increasing salience of the benefits of online grocery, modeling steps in behavior change, giving facts to address mistrust or improve control, asking questions to promote engagement, adding anonymized quotations from the pilot participants to reinforce social norms.
  Arms: Texting + Financial Incentive; Texting + Financial Incentive + Shoppable List; Texting + Shoppable List; Texting only
Behavioral: Financial incentive — Participants randomized to this component (alone or in combination with another experimental condition) will receive $1 for each dollar spent on fresh, frozen, or canned FVL loaded onto Instacart Fresh Funds, verified based on the submitted online grocery receipt or data from Instacart. The incentive applies to online purchases only and will not be earned for in-store transactions. A maximum weekly matched incentive will be set to $10, following the local FV incentive NYC ("Get the Good Stuff"). Fresh Funds earned, supported by Instacart Health, is an infrastructure integrated with retailer payment systems. Incentives will only be used for purchases of healthier foods (FVL) predetermined by the research team, as it has been used by FV prescription programs.
  Arms: Financial Incentive; Financial Incentive + Shoppable List; Texting + Financial Incentive; Texting + Financial Incentive + Shoppable List
Behavioral: Grocery list with instant shoppable SNAP-Ed recipes — Participants randomized to this component will receive weekly SNAP-Ed-based meal plans with instant shoppable grocery lists tailored to household size, dietary, and cultural preferences. All recipes will emphasize FVL-based eating patterns with Hispanic cuisine influences that have FVL as primary ingredients. Grocery lists organized by store department and recipe, will reflect the nearest available in-store unit. For example, if one recipe calls for 1 cup of flour, a small flour bag will be added to the list. Weekly meal plans will be shared via text as a photo and mailed as hard copies, with instant shoppable lists generated through Instacart's List feature as a hyperlink. Links to the instant shoppable list will be shared via text. Upon clicking, grocery items will be pre-filled automatically in the participant's online shopping cart. Participants can modify items and quantities before checking out.
  Arms: Financial Incentive + Shoppable List; Shoppable List; Texting + Financial Incentive + Shoppable List; Texting + Shoppable List

SUMMARY:
Food insecurity, that is, the lack of consistent access to nutritious and affordable food, is associated with poor diet, increased cardiovascular disease (CVD) risk, and has a negative long-term impact on the economy through increased health care costs. CVDs and food insecurity disproportionately affect Black and Hispanic families, and most of these racial health disparities can be attributed to social determinants of health, including poor access to healthy foods. A recent policy in the U.S. authorized the Supplemental Nutrition Assistance Program (SNAP) benefits to be used online to increase grocery access and promote healthy eating. Although online grocery shopping has been growing among populations of low-income, the selection of fruits, vegetables, and legumes (FVL), which are protective against CVD, is lower than in-store. Distrust of online hired shoppers' choices, fear of losing money on unsatisfactory purchases, and impulse of unhealthy food purchases have been the major barriers to online healthy food selection. Thus, there is a need for intervention packages that are effective, economical, and easily scalable into policies that address CVD-related outcomes and improve health equity. The proposed work will use a highly efficient methodological approach, the Multiphase Optimization Strategy (MOST), to test three experimental components aimed at barriers to online healthy food selection, called OPT-FRESH. This approach addresses weaknesses in prior studies, which cannot determine which elements of multicomponent interventions meaningfully improve outcomes. 360 families with children living in low-income urban communities of NYC will be randomized to receive some combination of the three experimental components for 12 weeks: 1) weekly text messages to improve the trust in online grocery services (off/on); 2) weekly match-up to $10 as a financial incentive for purchasing FVL online targeting loss aversion (off/on); 3) weekly instant shoppable grocery lists of culturally tailored meal suggestions using SNAP recipes targeted at impulse purchases (off/on). Delivery fee waiver and a tutorial video addressing digital literacy will be constant components to promote equity in participant enrollment. Aim 1 will determine the combination(s) of the three experimental components that improve overall household FVL purchase and food insecurity (primary outcomes) and FVL intake of children (secondary outcome). Aim 2 will identify the optimized intervention that balances component(s) that are affordable and scalable (high adoption, implementation, maintenance) that still produce meaningful effects on the outcomes, using decision analysis for intervention value efficiency. Aim 3 will determine the mechanistic effects of the three intervention components on the outcomes using factorial mediation analysis. Working with community-based organizations and nutrition and hunger relief programs in NYC, a grocery delivery service, and a team with unparalleled expertise in experimental trials, policy, and MOST, we will implement optimized, affordable, and scalable intervention strategies to improve neighborhood food access and ultimately CVD outcomes in socially vulnerable families.

DETAILED DESCRIPTION:
OPT-FRESH will use a highly efficient methodological approach for intervention development, the multiphase optimization strategy (MOST). We will partner with the private sector (Instacart) to leverage strategies from the public sector (SNAP) and test three experimental components aimed at barriers to online healthy food selection. The three experimental components, which were found in our pilot work to be feasible and acceptable, include: 1) weekly text messages to improve trust in online grocery services; 2) weekly match of up to $10 as a financial incentive for purchasing FVL online; and 3) weekly instant shoppable grocery lists of tailored meal suggestions using SNAP-Ed recipes. Moreover, as our pilot demonstrated that waiving delivery fees enabled more equitable participant enrollment and online grocery uptake, all participants will have the online delivery fee waived for the intervention period (12 weeks), along with a tutorial video addressing digital literacy to further promote equity in enrollment. A sample of 360 families with young children living in low-income urban communities of NYC will be randomized to receive some combination of the experimental components for 12 weeks. We will test component effects at 12 weeks and test maintenance in the absence of intervention (no fee waiving, experimental components) 9 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 21 years old)
* Live in a household with a young child(ren) under the age of 10 years and above age 2.
* Primary shopper for the household
* Have access to a smartphone or computer to place online orders
* Participation in the Supplemental Nutrition Assistance Program in the past year or income eligible (annual household income =< 130% of the federal poverty line)
* Agree to share itemized grocery receipts during the study (12 months)
* Willing to order groceries online
* English or Spanish speaker
* Informed consent

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Household Food Security | 6 weeks, 12 weeks, and 12 months
  Change in household food security from baseline will be measured using the 18-item validated USDA screening tool mid-intervention (6-week), post-intervention (12-week), and maintenance (12 months)
Household Purchase of Fruit, Vegetable, and Legumes. | 6 weeks, 12 weeks, and 12 months
  Change in household purchase of fruits, vegetables, and legumes (online and in-store) from baseline will be assessed via itemized grocery receipts obtained via text messages mid-intervention (6-week), post-intervention (12-week), and maintenance (12 months)

SECONDARY OUTCOMES:
Consumption of Fruit, Vegetable, and Legumes | 12 weeks
  Change in consumption of fruits and vegetables from baseline will be assessed via skin carotenoid using Veggie Meter in-person among adults and children at baseline and at 12-week

OTHER OUTCOMES:
Consumption of Fruit and Vegetable, and Legumes | 12 weeks
  Change in dietary intake from baseline will be measured via Dietary Screener Questionnaire (DSQ) reported online at baseline and 12-weeks.
Body Mass Index | 12 weeks
  Change in Body Mass Index from baseline will be measured via a body weight scale and stadiometer in-person among adults and children at baseline and 12-week.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Trude, PhD, Principal Investigator — New York University

IPD SHARING:
Plan to Share IPD: No
At this time, there are no plans to share IPD due to limitations related to participant privacy, the sensitive nature of the data collected, and constraints in the informed consent process that do not allow for broad data sharing. While we support data transparency, any future sharing would require additional ethical review and participant re-consent to ensure privacy protections are upheld.

DOCUMENTS (2):
  • Informed Consent Form: Informed Consent Form (Caregivers) (2026-01-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT07071753/ICF_000.pdf
  • Informed Consent Form: Child Assent Form (Child age 2-10 years old) (2026-01-22): https://cdn.clinicaltrials.gov/large-docs/53/NCT07071753/ICF_001.pdf